CLINICAL TRIAL: NCT00482612
Title: A Two-Week, Double Blind, Placebo-Controlled, Randomized, Parallel Group, Efficacy and Safety Out-Patient Trial With Org 50081 in Patients With Chronic Primary Insomnia
Brief Title: Study of the Safety and Effectiveness of Esmirtazapine in Participants With Chronic Primary Insomnia (P05706)
Acronym: RUBY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05706; 176001 (Other: Protocol number); MK-8265-003 (Other: Protocol number)
Record Dates: First submitted 2007-06-01; First posted 2007-06-05 (Estimated); Results first posted 2014-07-10 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Esmirtazapine 1.5 mg (Experimental): Esmirtazapine 1.5 mg tablet, oral administration in the evening, once daily, for 2 weeks
  Interventions: Drug: Esmirtazapine
- Esmirtazapine 3.0 mg (Experimental): Esmirtazapine 3.0 mg tablet, oral administration in the evening, once daily, for 2 weeks
  Interventions: Drug: Esmirtazapine
- Esmirtazapine 4.5 mg (Experimental): Esmirtazapine 4.5 mg tablet, oral administration in the evening, once daily, for 2 weeks
  Interventions: Drug: Esmirtazapine
- Placebo (Placebo Comparator): Placebo to esmirtazapine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esmirtazapine — Esmirtazapine maleate was provided as tablets for oral use containing either 1.5, 3.0, or 4.5 mg of active compound. In addition, tablets contain the following excipients: hydroxypropyl cellulose, maize starch (United States Pharmacopeia [USP] name: corn starch), magnesium stearate, and lactose monohydrate. Tablets were administered orally once daily about 30 minutes prior to bedtime.
  Other Names: Org 50081; MK-8265
  Arms: Esmirtazapine 1.5 mg; Esmirtazapine 3.0 mg; Esmirtazapine 4.5 mg
Drug: Placebo — Placebo tablets containing the following excipients: hydroxypropyl cellulose, maize starch (USP name: corn starch), magnesium stearate, and lactose monohydrate. Tablets were administered orally once daily about 30 minutes prior to bedtime.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if esmirtazapine (Org 50081) is a safe and effective treatment for insomnia. It was anticipated that esmirtazapine would increase mean Total Sleep Time (TST) as recorded in sleep diaries relative to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Has signed written informed consent after the scope and nature of the investigation was explained to them
* Has difficulty falling asleep, maintaining sleep or has early morning awakenings

Exclusion Criteria:

* Significant medical or psychiatric illness causing sleep disturbances
* Has a history of bipolar disorder or family (immediate family) of suicide
* Has sleep disorder such as sleep related breathing disorder, restless leg syndrome, narcolepsy
* Has significant other medical illness such as acute or chronic pain, heart, kidney or liver disease within the last year
* Currently diagnosed or meets the criteria for Major Depressive Disorder (MDD) or has been treated for MDD with the last 2 years
* Substance abuse, excessive use of alcohol (as determined by the physician) or drug addiction within the last year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2006-12-07 (Actual); Primary Completion 2008-08-11 (Actual); Study Completion 2008-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ivgy-May N, Roth T, Ruwe F, Walsh J. Esmirtazapine in non-elderly adult patients with primary insomnia: efficacy and safety from a 2-week randomized outpatient trial. Sleep Med. 2015 Jul;16(7):831-7. doi: 10.1016/j.sleep.2015.03.005. Epub 2015 Mar 30. PMID 26047890

RESULTS

PARTICIPANT FLOW:
Groups:
- Esmirtazapine 1.5 mg: Participants took esmirtazapine 1.5 mg tablets once daily by mouth during the 14-day In-treatment Period. Participants were followed for safety during a Follow-up Period, in which no study medication was administered.
- Esmirtazapine 3.0 mg: Participants took esmirtazapine 3.0 mg tablets once daily by mouth during the 14-day In-treatment Period. Participants were followed for safety during a Follow-up Period, in which no study medication was administered.
- Esmirtazapine 4.5 mg: Participants took esmirtazapine 4.5 mg tablets once daily by mouth during the 14-day In-treatment Period. Participants were followed for safety during a Follow-up Period, in which no study medication was administered.
- Placebo: Participants took placebo tablets once daily by mouth during the 14-day In-treatment Period. Participants were followed for safety during a Follow-up Period, in which no study medication was administered.
Period: In-treatment Period
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Esmirtazapine 4.5 mg | Placebo
Started | 137 | 125 | 129 | 135
Treated | 137 | 125 | 128 | 135
Completed | 137 | 125 | 128 | 135
Not Completed | 0 | 0 | 1 | 0
Not completed — No study medication administered | 0 | 0 | 1 | 0
Period: Follow-up Period
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Esmirtazapine 4.5 mg | Placebo
Started | 137 | 125 | 128 | 135
Completed | 123 | 107 | 106 | 127
Not Completed | 14 | 18 | 22 | 8
Not completed — Other | 4 | 2 | 1 | 2
Not completed — Lack of compliance | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 4 | 2 | 1
Not completed — Adverse Event | 4 | 7 | 9 | 0
Not completed — Lack of Efficacy | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 5 | 7 | 2
Not completed — Reasons not related to trial | 1 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported for the All-Subjects-Treated group. One participant who was randomized to receive MK-8265 4.5 mg did not receive double-blind study medication.
Groups:
- Esmirtazapine 1.5 mg: Participants took esmirtazapine 1.5 mg tablets once daily by mouth during the 14-day In-treatment Period. No study medication was administered during the Follow-up Period.
- Esmirtazapine 3.0 mg: Participants took esmirtazapine 3.0 mg tablets once daily by mouth during the 14-day In-treatment Period. No study medication was administered during the Follow-up Period.
- Esmirtazapine 4.5 mg: Participants took esmirtazapine 4.5 mg tablets once daily by mouth during the 14-day In-treatment Period. No study medication was administered during the Follow-up Period.
- Placebo: Participants took placebo tablets once daily by mouth during the 14-day In-treatment Period. No study medication was administered during the Follow-up Period.
- Total: Total of all reporting groups
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Esmirtazapine 4.5 mg | Placebo | Total
Number analyzed (Participants) | 137 | 125 | 128 | 135 | 525
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.8 (12.4) | 45.6 (12.0) | 44.5 (12.2) | 46.2 (11.3) | 45.3 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 85 | 72 | 90 | 339
  Male | 45 | 40 | 56 | 45 | 186

OUTCOME MEASURES:

1. Primary Outcome: Average Total Sleep Time (TST) as Recorded Daily in the Sleep Diary During the 14-day In-treatment Period
Description: TST was defined as the total amount of time (measured in minutes) that was actually spent sleeping the previous night as recorded daily in the participant's sleep diary. TST values over the 14-day active treatment period were averaged for each participant, and average TST was then reported by treatment arm. For participants with missing data, the average of the nights for which TST data were present was used in the analysis.
Time Frame: Day 1 to Day 15
Population: The Intent-To-Treat Group consisted of all randomized participants who received at least one dose of double-blind trial medication, and had baseline and at least one post-baseline measurement for at least one efficacy assessment.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Esmirtazapine 1.5 mg: Participants took esmirtazapine 1.5 mg tablets once daily by mouth during the 14-day In-treatment Period.
- Esmirtazapine 3.0 mg: Participants took esmirtazapine 3.0 mg tablets once daily by mouth during the 14-day In-treatment Period.
- Esmirtazapine 4.5 mg: Participants took esmirtazapine 4.5 mg tablets once daily by mouth during the 14-day In-treatment Period.
- Placebo: Participants took placebo tablets once daily by mouth during the 14-day In-treatment Period.
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Esmirtazapine 4.5 mg | Placebo
Number analyzed (Participants) | 135 | 121 | 126 | 133
Minutes | 382.14 (68.155) | 382.77 (81.172) | 394.83 (85.575) | 351.40 (78.551)
Statistical Analysis 1: Comparison: Esmirtazapine 1.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Baseline TST was used as a covariate
Statistical Analysis 2: Comparison: Esmirtazapine 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Baseline TST was used as a covariate
Statistical Analysis 3: Comparison: Esmirtazapine 4.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Baseline TST was used as a covariate

2. Secondary Outcome: Average Sleep Latency (SL) as Recorded Daily in the Sleep Diary During the 14-day In-treatment Period
Description: SL was defined as the duration of time measured in minutes that it took a participant to fall asleep as recorded daily in the participant's sleep diary. SL values over the 14-day active treatment period were averaged for each participant, and average SL was then reported by treatment arm. For participants with missing data, the average of the nights for which TST data were present were used in the analysis.
Time Frame: Day 1 to Day 15
Population: The Intent-To-Treat Group consisted of all randomized participants who received at least one dose of double-blind trial medication and had baseline and at least one post-baseline measurement for at least one efficacy assessment.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Esmirtazapine 4.5 mg | Placebo
Number analyzed (Participants) | 135 | 121 | 126 | 133
Minutes | 48.93 (34.59) | 52.02 (38.95) | 50.80 (45.76) | 60.13 (42.98)
Statistical Analysis 1: Comparison: Esmirtazapine 1.5 mg vs Placebo; Test type: Superiority or Other; p = 0.0014, ANCOVA; Baseline SL was used as a covariate
Statistical Analysis 2: Comparison: Esmirtazapine 3.0 mg vs Placebo; Test type: Superiority or Other; p = 0.0135, ANCOVA; Baseline SL was used as a covariate
Statistical Analysis 3: Comparison: Esmirtazapine 4.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Baseline SL was used as a covariate

3. Secondary Outcome: Number of Participants Experiencing an Adverse Event (AE) During the 14-day In-treatment Period
Description: The total number of participants with an AE during the 14-day In-treatment Period was tallied for each treatment arm. An AE was defined as any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: Day 1 to Day 15
Population: The All-Subjects-Treated Group consisted of all participants who received at least 1 dose of trial medication.
Measure: Number; unit: Number of participants
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Esmirtazapine 4.5 mg | Placebo
Number analyzed (Participants) | 137 | 125 | 128 | 135
Number of participants | 35 | 41 | 41 | 28

4. Secondary Outcome: Number of Participants Who Discontinued From Study Treatment Due to an AE During the 14-day In-Treatment Period
Description: The total number of participants discontinuing from study treatment due to experiencing an AE was tallied for each treatment arm. An AE was defined as any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: Day 1 to Day 15
Population: The All-Subjects-Treated Group consisted of all participants who received at least 1 dose of trial medication.
Measure: Number; unit: Number of participants
Arm/Group | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Esmirtazapine 4.5 mg | Placebo
Number analyzed (Participants) | 137 | 125 | 128 | 135
Number of participants | 4 | 7 | 9 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 of the Treatment Period up to 30 days after completion of the Treatment Period (up to 45 days). AE data were not reported for the 1 enrolled participant who did not receive study medication.
Description: AEs were collected for 525 treated participants separately during the In-Treatment Period (Days 1-15) and during the Follow-up Period (up to Day 45).
Groups:
- Esmirtazapine 1.5 mg In-treatment: Participants took esmirtazapine 1.5 mg tablets once daily by mouth during the 14-day In-treatment Period.
- Esmirtazapine 3.0 mg In-Treatment: Participants took esmirtazapine 3.0 mg tablets once daily by mouth during the 14-day In-treatment Period.
- Esmirtazapine 4.5 mg In-treatment: Participants took esmirtazapine 4.5 mg tablets once daily by mouth during the 14-day In-treatment Period.
- Placebo In-treatment: Participants took placebo tablets once daily by mouth during the 14-day In-treatment Period.
- Esmirtazapine 1.5 mg Follow-up: After receiving 1.5 mg esmirtazipine in the In-Treatment Period, participants were followed for safety during a Follow-up Period in which no study medication was administered.
- Esmirtazapine 3.0 mg Folow-up: After receiving 3.0 mg esmirtazipine in the In-Treatment Period, participants were followed for safety during a Follow-up Period in which no study medication was administered.
- Esmirtazapine 4.5 mg Follow-up: After receiving 4.5 mg esmirtazipine in the In-Treatment Period, participants were followed for safety during a Follow-up Period in which no study medication was administered.
- Placebo Follow-up: After receiving placebo in the In-Treatment Period, participants were followed for safety during a Follow-up Period in which no study medication was administered.
Arm/Group | Esmirtazapine 1.5 mg In-treatment | Esmirtazapine 3.0 mg In-Treatment | Esmirtazapine 4.5 mg In-treatment | Placebo In-treatment | Esmirtazapine 1.5 mg Follow-up | Esmirtazapine 3.0 mg Folow-up | Esmirtazapine 4.5 mg Follow-up | Placebo Follow-up
Serious Adverse Events (participants affected / at risk) | 2/137 | 1/125 | 1/128 | 0/135 | 0/137 | 0/125 | 0/128 | 0/135
Other Adverse Events (participants affected / at risk) | 10/137 | 11/125 | 9/128 | 2/135 | 0/137 | 0/125 | 0/128 | 0/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esmirtazapine 1.5 mg In-treatment (N=137) | Esmirtazapine 3.0 mg In-Treatment (N=125) | Esmirtazapine 4.5 mg In-treatment (N=128) | Placebo In-treatment (N=135) | Esmirtazapine 1.5 mg Follow-up (N=137) | Esmirtazapine 3.0 mg Folow-up (N=125) | Esmirtazapine 4.5 mg Follow-up (N=128) | Placebo Follow-up (N=135)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominoplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esmirtazapine 1.5 mg In-treatment (N=137) | Esmirtazapine 3.0 mg In-Treatment (N=125) | Esmirtazapine 4.5 mg In-treatment (N=128) | Placebo In-treatment (N=135) | Esmirtazapine 1.5 mg Follow-up (N=137) | Esmirtazapine 3.0 mg Folow-up (N=125) | Esmirtazapine 4.5 mg Follow-up (N=128) | Placebo Follow-up (N=135)
Somnolence (Nervous system disorders) | 10 (10) | 11 (11) | 9 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications must be based on data validated and released by the Sponsor. Any such scientific paper, presentation, or other communication concerning the clinical trial will first be submitted to the Sponsor, at least 6 weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.